CLINICAL TRIAL: NCT02502591
Title: Pudendal Nerve Block for Postoperative Pain Relief in Women Undergoing Posterior Vaginal Repairs: a Pilot Study
Brief Title: Pudendal Nerve Block for Postoperative Posterior Repair Pain Relief
Acronym: PPPR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1510152
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2017-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Additional pain relief (a Pudendal Nerve Block (PNB)) will be administered during surgery in addition to routine care.
  Interventions: Drug: Pudendal Nerve Block
- control (No Intervention): routine care only

INTERVENTIONS:
Drug: Pudendal Nerve Block — An injection of local anaesthetic (3 ml of 0.25% bupivacaine) will be administered around the trunk of the pudendal nerve.
  Other Names: PNB
  Arms: intervention

SUMMARY:
Rectocoele or a posterior vaginal prolapse (bulge in the vagina) is a frequent gynaecological condition. It is repaired by repairing and reinforcing the support to the vaginal wall at the back. A small cut is made through the lining of the back wall of the vagina. The supports to the rectum are reinforced with stitches and the bulging part of the vaginal wall cut away. The wound in the vagina is then stitched up. Rectocoele repair is usually carried under a general anaesthetic with women reporting moderate to severe degrees of pain post operatively on sitting down.

A Pudendal Nerve Block (PNB) is a common analgesic (pain killing) technique often used for women who need an instrumental delivery during childbirth. It is also widely used during a range of surgical procedures (operations) as a preventive analgesia to help reducing post -operative pain. The investigators would like to see if using this technique during routine rectocele repair will help with post - op pain.

DETAILED DESCRIPTION:
Pelvic Organ Prolapse (POP) can occur in up to 50% of women after childbirth. Common complications include urinary infection, postoperative pain, and wound infection.

The majority of prolapse repair procedures are carried out under general anaesthetic (GA) with regular analgesia required post operatively. The pain is often described as "agonizing" and results in a substantial consumption of analgesia, often leading to extended periods of bladder catheterisation and bowel dysfunction. Despite numerous attempts to modify surgical techniques and anaesthetic regimens, the problems persist.

In an attempt to relieve the problem local clinicians have had promising results from the addition of a standardised preventive Pudendal Nerve Block (PNB) in reducing post- op pain. To widen the clinical utility of this procedure an evidence base will be required.

Preventive analgesia: Preventive analgesia is a broad term used to describe an analgesic regime given during surgery to control post - op pain and its aim is to reduce the impact of the process known as central sensitization. This refers to an increase in synaptic efficacy in the somatosensory neurons following tissue injury (e.g. surgery) or nerve damage. This leads to a reduction in pain threshold, an amplification of pain responses and a spread of pain sensitivity to non-injured areas resulting in increased post -op pain intensity and analgesic requirements. Preventive analgesics (including nerve blocks) have been incorporated into a range of surgical procedures, with a recent review identifying its strong positive impact on post-operative pain and analgesic consumption.

The Pudendal nerve is a mixed nerve (sensory and motor) derived from the somatic component of sacral nerve roots S2-S4. It is located behind the sacrospinous ligament. It supplies anal and urethral sphincters, the pelvic floor muscles, anal and perineal skin. PNB is a routine procedure used during instrumental deliveries in obstetrics and as a low-risk, low-cost anaesthetic technique effectively reducing perineal and vaginal discomfort during repair of obstetric lacerations. PNB is also increasingly being utilised as a preventive analgesia with positive results on pain relief, reduced analgesics, improved spontaneous micturition, less pain on defecation and shorter hospital stay and pain on following haemorrhoidectomy. Improving post- operative pain relief and enhancing patient recovery is of fundamental importance to both the individual and the National Health Service (NHS). This study is a preliminary step in the assessment of a preventive analgesia on women's post- op experience following routine posterior vaginal wall surgery.

Hypothesis: The addition of a PN), administered during routine rectocele repair being carried out under general anaesthetic (GA), will provide more effective and prolonged postoperative analgesia and shorter hospital stay compared to receiving GA alone.

Aim: To obtain preliminary data on the impact of administering a standard PNB during routine rectocele repair on women's post-op experience, and assess the feasibility of future studies on the potential for the procedure to become a routine part of clinical practice.

Objectives are to assess: the feasibility of recruitment and retention, the impact of the PNB on women's post-op experience, and obtain preliminary data to inform sample size calculations and refine outcome measures for future studies.

Study design: This is a pilot/feasibility study being undertaken within the Gynaecology Department of the Royal Devon and Exeter NHS Foundation Trust (RD&E NHS FT).

Recruitment: It is anticipated that potential participants will be identified from routine clinical care, with clinicians informing patients of the project in general terms and seeking permission for their contact details to be passed to the research team. Potential participants will then be contacted by a member of the research team and given more detailed verbal and written information. This will then be followed by a further opportunity for discussion with the research team prior to being invited to participate in the study.

All potential participants who fulfil the entry criteria will be invited to take part. This will enable a realistic assessment of recruitment and the recruitment strategy.

Procedure: Written informed consent will be obtained prior to any study procedures. This will include permission to access routinely collected data from the participant's medical notes.

Baseline data will include: height, weight, and current medicines (including routine analgesia). Participants will be randomised to either the intervention group (General Anaesthetic (GA) and PNB) or control group (GA alone) by a computer generated randomisation schedule.

Surgical procedure: Participants will undergo routine posterior vaginal wall surgery following standard surgical procedures and protocols.

For those randomised to the intervention group - a standardised PNB will be administered prior to completion of surgery.

Standardised PNB: A PNB will be performed by injection of local anaesthetic around the trunk of the pudendal nerve, which is located behind the sacrospinous ligament. Using transvaginal approach, the ischial spines will be palpated posterolateral to the vaginal sidewall. The sacrospinous ligament is a firm band running medially and posteriorly from the ischial spine to the sacrum. The needle guide with the needle and syringe containing anaesthetic will be inserted so the tip lies against the vaginal mucosa about 1 cm medial and posterior to the ischial spine. When the needle guide gets properly positioned, the needle will be pushed beyond its tip and through the vaginal mucosa into the sacrospinous ligament. After aspirating to confirm the absence of an intravascular location, 3 ml of 0.25% bupivacaine will be injected into the ligament. The needle will then be advanced slightly until the sensation of resistance caused by the ligament is lost. The needle has to be lodged in the loose areolar tissue behind the ligament where the pudendal nerve will be located. Aspiration will again be performed to confirm the absence of an intravascular position (the pudendal and inferior gluteal vessels lie adjacent to the pudendal nerve), and then the remaining 7 mL of anaesthetic are injected. The procedure will be repeated on the contralateral side.

Post -op: For all participants the investigators will record: post -operative pain (Visual Analogue Scale (VAS) score) at 6, 12, 24, 36 and 48 hours, length of bladder catheterisation, pain associated with defecation and analgesic consumption.

Data Collection and Recording: All participants will be assigned a unique study identifier (ID) All data collected will be recorded and stored under this ID number. Data will be initially recorded onto a study specific data collection form (DCF). Data will then be recorded onto a study specific database. Hard/scanned copies will be stored in the study specific site file. To ensure data quality, data collected and recorded will be screened and reviewed for discrepancies and missing data prior to analysis.

Confidentiality: data will be held in a link-anonymised format, with personal identifiable data only accessible to personnel with training in data protection. Participants' research and sample data will be identified by unique study ID numbers and all data will be held on password-protected computers Data Storage and Archiving: All consent and paper data collection forms will be scanned onto discs and stored in a locked filing cabinet within the CI's controlled access office in the Centre for Women's Health for the duration of the project. Paper copies will be shredded. At the end of the project, all study data will be archived as per standard Research and Development (R&D) department protocol.

Primary Outcome measure: Post- op pain scores as defined by VAS measure Secondary outcome measures: Length of bladder catheterisation, pain associated with defecation and post-op analgesic consumption Statistics and Power Calculations: The aim of this study is to obtain preliminary data and determine the feasibility of a future Randomised Control Trial (RCT), not to determine clinical differences. The investigators estimate 40 potential participants will be available over a 9 month period (figures obtained from RD&E Gynaecology Surgery dept. based on last year's operation lists). The investigators will invite all patients who fulfil the entry criteria to participate. This will enable us to determine a realistic recruitment rate and obtain estimates of differences in post-op pain scores to inform a full RCT. Analysis will be restricted to descriptive statistics only.

Adverse events/patient safety: It is not anticipated that participants involved in this project will be subject to adverse effects. Pudendal Nerve blocks are very rarely associated with complications such as anaphylaxis, haematoma and infection at the site of injection, ischial paraesthesias and systemic toxicity due to intravascular administration. The risk of these rare complications would apply to any nerve block currently used in routine clinical practice. The risks will be further minimised by the procedure being carried out by a Gynaecological Consultant experienced in the procedure, with full anaesthetic and surgical team back up if required. The CI will be informed of any adverse effects within 24 hours and they will be reported following local NHS R&D protocols, with a copy of any adverse event form stored in the project site file.

Subjects will be informed that they are free to withdraw from the study at any time up until their data are coded but not anonymised. When data are fully anonymised, the participants will still be able to withdraw but their data will be retained.

During routine clinical care the clinicians involved with the study have had in-depth discussions with the women in their care including treatment options and the potential complications associated with surgery. Of particular concern to patients is how much pain they will be in, leading to the initial idea of the use of PNB to relieve post-op pain. Resultant anecdotal feedback suggested this resulted in lower post-op pain levels than other patients in the ward that had similar operations. This led directly to the development of the current project.

The investigators subsequently discussed the proposal with a cross section of women attending the pre- and post op Pelvic Organ Prolapse (POP) clinics. All expressed enthusiasm for the project and a willingness to be involved either as a participant or as a user representative on any further definitive studies.

Blinding: on recruitment, a member of the clinical surgical team (not a member of the research team) will open the next in line randomisation envelope and identify to the surgeon the participant's group allocation. This will then be recorded against the participant's unique study ID.

Un-blinding: Should a serious, adverse event or clinical situation occur that required a participant to be un-blinded, that decision will be made by the Chief Investigator (CI) and reported to the sponsor as per standard R&D Dept. Governance protocol? Time scale: 12 months. In the short term the study will provide preliminary data to on the impact of administering a PNB to women undergoing routine posterior vaginal wall surgery. In the longer term this data will inform a future definitive study into the clinical and economic impact of the routine use of PNB in this context. Results will be written up and submitted for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing isolated posterior vaginal wall repair under GA
* Age 20-80 yrs
* Wiling and able to provide informed consent

Exclusion Criteria:

* Women undergoing concomitant anterior repairs, vaginal hysterectomies or mesh repair
* History of chronic pelvic pain.
* Known allergy to local anaesthetic agents
* Unable/unwilling to provided informed consent

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Post- op pain scores. as defined by VAS measure | over a 48 hour post-operative period.
  Pain score defined by Visual Analogue Scores (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Kay, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- NIHR Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No